CLINICAL TRIAL: NCT02615691
Title: Phase 3, Prospective, Multi-center, Open Label Study to Investigate Safety, Immunogenicity and Hemostatic Efficacy of PEGylated Factor VIII (BAX 855) in Previously Untreated Patients (PUPs) < 6 Years With Severe Hemophilia A (FVIII < 1%)
Brief Title: A Study of PEGylated Recombinant Factor VIII (BAX855) in Previously Untreated Young Children With Severe Hemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 261203; 2015-002136-40 (EudraCT Number)
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — BAX 855

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): Previously Untreated Patients (PUPs) < 6 years of age with severe hemophilia A (FVIII < 1%) and < 3 exposure days (EDs) to ADVATE, BAX 855 or plasma transfusion were enrolled in a single arm group.
  Part A (Main Study): Participants age <3 years - who had not experienced two joint bleeds received on-demand treatment of 10-80 international units per kilogram (IU/kg) intravenously (IV) depending on the severity of the bleeding episode; and - who experienced maximum of two joint bleeds received prophylaxis treatment with dose of 25-80 IU/kg of BAX 855 IV (based on investigator discretion) once weekly for up to 100 EDs.
  Part B (Immune tolerance induction [ITI] Portion): Participants who met the pre-defined Part B treatment criteria entered Part B of the study for ITI. Participants either received prophylaxis treatment of BAX 855 low dose 50 IU/kg IV, three times a week or high dose 100-200 IU/kg IV, daily at discretion of the investigator according to the institution's standard of care.
  Interventions: Biological: PEGylated Recombinant Factor VIII; Biological: ITI

INTERVENTIONS:
Biological: PEGylated Recombinant Factor VIII — Polyethylene glycol (PEG)-ylated full-length recombinant FVIII (rFVIII).
  Other Names: ADYNOVATE; BAX 855; TAK-660
Biological: ITI — Immune tolerance induction therapy

SUMMARY:
This study is for young children with severe hemophilia A who have previously not been treated with BAX855 or other FVIII concentrates.

The main aim of the study is to check for side effects from treatment with BAX855. This includes the buildup of antibodies against FVIII which may stop BAX855 from working properly. Another aim is to learn how well BAX855 controls bleeding.

In this study, the children can receive BAX855 either as preventative treatment (prophylaxis), or as needed to treat bleeding (on-demand).

In case a participant develops antibodies, treatment will be provided as part of the study.

ELIGIBILITY:
Inclusion Criteria

1. Participant is <6 years old at the time of screening.
2. Participant is previously untreated with <3 exposure days (EDs) to ADVATE, BAX 855 or plasma transfusion at any time prior to screening.
3. Participant has severe hemophilia A (Factor VIII (FVIII) <1%) as determined by the central laboratory, or a historical FVIII level <1% as determined at any local laboratory, optionally supported by an additional FVIII gene mutation consistent with severe hemophilia A.
4. Participant is immune competent with a cluster of differentiation 4 (CD4+) count > 200 cells per cubic millimeter (mm^3), as confirmed by the central laboratory at screening.
5. Parent or legally authorized representative is willing and able to comply with the requirements of the protocol.

Additional inclusion criteria for Part B (immune tolerance induction [ITI]).

1. Parent or legal representative has/have voluntarily provided signed informed consent for ITI portion.
2. Participant has a confirmed positive high titer inhibitor (> 5.00 Bethesda unit (BU)) or has a positive confirmed low titer inhibitor (greater than or equal to [>=] 0.6 BU) as determined by the central laboratory based on a second repeat blood sample with

   1. poorly controlled bleeding despite increased BAX 855 doses, or
   2. requires bypassing agents to treat bleeding.

Exclusion Criteria

1. Participant has detectable FVIII inhibitory antibodies (>=0.6 BU using the Nijmegen modification of the Bethesda assay) as confirmed by central laboratory at screening.
2. Participant has a history of FVIII inhibitory antibodies (>=0.6 BU using the Nijmegen modification of the Bethesda assay or the Bethesda assay) at any time prior to screening.
3. Participant has been diagnosed with an inherited or acquired hemostatic defect other than hemophilia A (eg, qualitative platelet defect or von Willebrand's disease).
4. Participant has been previously treated with any type of FVIII concentrate other than ADVATE or BAX 855, or was administered ADVATE, BAX 855 or plasma transfusion for >=3 EDs at any time prior to screening.
5. Participant receives > two EDs of ADVATE in total during the periods prior to enrollment and during the screening period, until the baseline infusion.
6. The participant's weight is anticipated to be <5 kilogram (kg) at the baseline visit.
7. Participant's platelet count is <100,000 per milliliter (mL).
8. Participant has known hypersensitivity towards mouse or hamster proteins, polyethylene glycol (PEG) or Tween 80.
9. Participant has severe chronic hepatic dysfunction (eg, >5 times upper limit of normal alanine aminotransferase [ALT], aspartate aminotransferase [AST], or a documented international normalized ratio [INR] >1.5) in his medical history or at the time of screening.
10. Participant has severe renal impairment (serum creatinine >1.5 times the upper limit of normal).
11. Participant has current or recent (<30 days) use of other PEGylated drugs prior to study participation or is scheduled to use such drugs during study participation.
12. Participant is scheduled to receive during the course of the study a systemic immunomodulating drug (e.g. corticosteroid agents at a dose equivalent to hydrocortisone greater than 10 mg/day or α-interferon) other than anti-retroviral chemotherapy.
13. Participant has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
14. Parent or legally authorized representative has a medical, psychiatric, or cognitive illness or recreational drug/alcohol use that, in the opinion of the investigator, would affect participant safety or compliance.
15. Parent, legally authorized representative or participant are a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie, children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study.

Additional exclusion criteria for Part B (ITI)

1. Spontaneous disappearance of the inhibitor prior to ITI.
2. FVIII inhibitor titer >=0.6 BU is not confirmed by a second new blood sample and determined at the central laboratory.
3. Inability or unwillingness to comply with the protocol.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (91):
- United States (20):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Kaiser Permanente Oakland M.C., Cupertino, California
  - Kaiser Permanente Oakland M.C., Oakland, California
  - Kaiser Permanente Oakland M.C., Roseville, California
  - UC Davis Health System, Sacramento, California
  - Connecticut Children's Med Ctr, Hartford, Connecticut
  - Univ Florida College Medicine, Gainesville, Florida
  - Center for Advanced Pediatrics, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's H, Chicago, Illinois
  - Bleeding and Clotting Dis.Inst., Peoria, Illinois
  - UMHS, Ann Arbor, Michigan
  - New York Presbyterian Hospital, New York, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Rainbow Babies/Childrens Htl, Cleveland, Ohio
  - Penn State MS Hershey Med Ctr, Hershey, Pennsylvania
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
- Medizinische Universitat Wien, Vienna, Austria
- Belgium (4):
  - HUDERF, Brussels
  - Cliniques Uni Saint-Luc, Brussels
  - Univ. Ziekenhuis Gent Apotheek, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
- Bulgaria (3):
  - UMHAT Sv. Georgi, EAD, Plovdiv
  - SHAT Oncohaematology Diseases, Sofia
  - MHAT Sv. Marina, EAD, Varna
- Canada (2):
  - Kaye Edmonton Clinic, Edmonton, Alberta
  - McMaster Health Science, Hamilton, Ontario
- Rigshospitalet Copenhagen, Copenhagen, Denmark
- Helsinki Univ Hospital, Helsinki, Finland
- France (5):
  - CHU CAEN Hopital Cote de Nacre, Caen, Calvados
  - Essais cliniques CHU Rennes, Rennes, Ille Et Vilaine
  - Hopital Necker Enfants Malades, Paris, Paris
  - Hopital Jeanne de Flandre - CHU Lille, Lille
  - CHU de Rouen, Rouen
- Germany (4):
  - Werlhof-Institut GmbH, Hanover, Lower Saxony
  - Inst. f. Experimentelle, Bonn
  - Klinik F.Haematologie,Onkologie, Düsseldorf
  - Poliklinik PaediaHaematologie, Hamburg
- Hong Kong (2):
  - The University of Hong Kong Queen Mary Hospital, Hong Kong
  - Chinese University Of Hong Kong, Shatin
- Hungary (2):
  - Belgyogyaszat Onkohaematologia, Budapest
  - Debreceni Egyetem, Debrece
- Italy (4):
  - Presidio Ospedaliero F. Alessi, Catania
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale Maggiore Policlinico, Milan
  - Umberto I Pol. di Roma-Università di Roma La Sapienza, Rome
- Malaysia (6):
  - Hospital Ampang, Ampang, Kuala Lumpur
  - Hospital HRPB, Ipoh, Perak
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching
  - Hospital Sultanah Nur Zahirah, Terengganu
- Universitair Medisch Centrum Groningen (UMCG), Groningen, Netherlands
- Oslo Universitetssykehus - Rikshospitalet, Oslo, Norway
- Singapore (2):
  - NUS YLL School of Medicine, Singapore
  - KKH, Singapore
- South Korea (4):
  - Eulji University Hospital, Daejeon
  - Severance Hospital, Yonsei, Seoul
  - Kyung Hee University Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (4):
  - Hospital Univ. Son Espases, Palma de Mallorca, Balearic Islands
  - HOSPITAL A Coruna, A Coruña
  - Hospital Universitario La Paz, Madrid
  - Hospital Univ del Rio Hortega, Valladolid
- Taiwan (4):
  - Kaohsiung Chung- Ho Memorial Hosp, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General, Taichung
  - Tri-Service General Hospital, Taipei
- Thailand (5):
  - Siriraj Hospital, Bangkoknoi, Bangkok
  - King Chulalongkorn Memorial, Patumwan, Bangkok
  - Ramathibodi Hospital, Ratchathewi, Bangkok
  - Srinagarind Hospital, Muang, Changwat Khon Kaen
  - Maharaj Nakorn Chiang Mai, Muang, Chiang Mai
- Turkey (Türkiye) (8):
  - Acibadem Adana Hospital, Adana
  - Hacettepe Üniversitesi, Ankara
  - Akdeniz Universitesi, Antalya
  - Uludag Universitesi Tip Fakültesi, Bursa
  - Istanbul Üniversitesi Cerrahpaşa, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
  - Erciyes Univers Tip Fakultesi, Kayseri
  - 19 Mayis Universitesi, Samsun
- Ukraine (3):
  - MI Cherkasy Reg Onc Dis of CRC, Cherkasy
  - SI Institute of Blood Pathology and Transfusion Medicine of NAMSU, Lviv
  - CI Zaporizhzhia Reg CCH of ZRC, Zaporizhzhia
- United Kingdom (4):
  - Royal Manchester Children's Hospital, Manchester, Greater Manchester
  - Univ Hospital Southampton, Southampton, Hampshire
  - Bristol Royal H. for Children, Bristol
  - Evelina Children's Hospital - St Thomas' Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda

REFERENCES:
- [Derived] Sidonio RF Jr, Thompson AA, Peyvandi F, Stasyshyn O, Yeoh SL, Sosothikul D, Antmen AB, Maggiore C, Engl W, Ewenstein B, Tangada S. Immunogenicity, safety, and efficacy of rurioctocog alfa pegol in previously untreated patients with severe hemophilia A: interim results from a phase 3, prospective, multicenter, open-label study. Expert Rev Hematol. 2023 Jul-Dec;16(10):793-801. doi: 10.1080/17474086.2023.2247160. Epub 2023 Sep 7. PMID 37646148
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc74db2bf003ab45e99

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites globally from 12 November 2015 to 29 October 2024.
Pre-assignment Details: Previously untreated patients (PUPs) <6 years with severe hemophilia A (Factor VIII [FVIII] <1%) were treated with BAX 855 in Part A of this study for at least 100 exposure days (EDs) or until they had developed a confirmed FVIII inhibitor. Then, participants who developed high or low titer FVIII inhibitors entered Part B. In Part B they underwent immune tolerance induction (ITI) with BAX 855.
Groups:
- All Participants: PUPs < 6 years of age with severe hemophilia A (FVIII < 1%) and < 3 EDs to ADVATE, BAX 855 or plasma transfusion were enrolled in a single arm group.
  Part A (Main Study): Participants age <3 years - who had not experienced two joint bleeds received on-demand treatment of 10-80 international units per kilogram (IU/kg) intravenously (IV) depending on the severity of the bleeding episode; and - who experienced maximum of two joint bleeds received prophylaxis treatment with dose of 25-80 IU/kg of BAX 855 IV (based on investigator discretion) once weekly for up to 100 EDs.
  Part B (ITI Portion): Participants who met the pre-defined Part B treatment criteria entered Part B of the study for ITI. Participants either received prophylaxis treatment of BAX 855 low dose 50 IU/kg IV, three times a week or high dose 100-200 IU/kg IV, daily at the discretion of the investigator according to the institution's standard of care.
Period: Part A: Main Study (5 Years)
Arm/Group | All Participants
Started | 120
Part A: On-demand Treatment (Participants who received at least one on-demand treatment of BAX 855 in Part A of the study. A participant that received on-demand treatment first and then moved to prophylaxis treatment was counted for both on-demand and prophylaxis regimens. A participant that started with prophylaxis treatment was counted only for the prophylaxis regimen even if the participant received on-demand treatment while on the prophylaxis regimen.) | 80
Part A: Prophylaxis Treatment (Participants who received at least one prophylaxis treatment of BAX 855 in Part A of the study.) | 112
Completed | 106
Not Completed | 14
Not completed — Adverse Event | 3
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 7
Not completed — Reason Not Specified | 2
Period: Part B: ITI Portion (3.5 Years)
Arm/Group | All Participants
Started | 7
Part B:FVII Inhibitor Treatment(50IU/kg 3 Times Weekly Regimen) (Participants received prophylaxis treatment of 50 IU/kg BAX 855 three times a week in Part B of the study.) | 4
Part B:FVII Inhibitor Treatment (100-200IU/kg Daily Regimen) (Participants received prophylaxis treatment of 100-200 IU/kg BAX 855 daily in Part B of the study.) | 3
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAS) included all participants in the enrolled population with at least one BAX 855 infusion.
Arm/Group | All Participants
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.90 (0.717)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 114
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 45
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 61
  More than one race | 4
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With FVIII Inhibitor Development
Description: Number of participants who developed an inhibitor (at any time) confirmed by a central laboratory based on a second repeat blood sample draw within 2 weeks of site notification of an inhibitor and all participants who had not developed an inhibitor and had greater than or equal to (>=) 100 EDs when the sample for the last valid inhibitor test was drawn.
Time Frame: Throughout Part A of the study, approximately 5 years
Population: The SAS included all participants in the enrolled population with at least one BAX 855 infusion. Included in the analysis were participants who had equal or greater than 100 EDs or developed a confirmed FVIII inhibitor.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Main Study: Participants age <3 years - who had not experienced two joint bleeds received on-demand treatment of 10-80 IU/kg IV depending on the severity of the bleeding episode; and - who experienced maximum of two joint bleeds received prophylaxis treatment with dose of 25-80 IU/kg of BAX 855 IV (based on investigator discretion) once weekly for up to 100 EDs.
Arm/Group | Part A: Main Study
Number analyzed (Participants) | 100
Participants | 11

2. Primary Outcome: Number of Participants With Success of Immune Tolerance Induction (ITI)
Description: Success is defined as 1) a persistently negative inhibitor titer less than (<) 0.6 Bethesda unit (BU), 2) FVIII IR >=66% of the baseline value following a wash-out period of 84-96 hours, and 3) a FVIII half-life of >=6 hours.
Time Frame: Up to 33 months in Part B of the study
Population: The FVIII Inhibitor Treatment Analysis Set (IAS) included all participants who received at least one FVIII inhibitor treatment with BAX 855 during the study after the date that participant moved to FVIII inhibitor treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: ITI Portion: Participants who met the pre-defined Part B treatment criteria entered in the Part B of the study for ITI. Participants either received prophylaxis treatment of low dose BAX 855 50 IU/kg IV, three times a week or high dose 100-200 IU/kg IV, daily at the discretion of the investigator according to the institution's standard of care.
Arm/Group | Part B: ITI Portion
Number analyzed (Participants) | 7
Participants | 5

3. Secondary Outcome: Number of Participants With Binding Immunoglobulin G (IgG) and Immunoglobulin M (IgM) Antibodies
Description: Binding IgG and IgM antibodies to FVIII , Factor VIII-Polyethylene glycol (PEG-FVIII) and Polyethylene glycol (PEG) was assessed. A participant that received on-demand treatment first and then moved to prophylaxis treatment was counted for both on-demand and prophylaxis regimens. A participant that started with prophylaxis treatment was counted only for the prophylaxis regimen even if the participant received on-demand treatment while on the prophylaxis regimen. Visits and their approximate time in weeks after baseline visit for individual participants: Visit 1(Week 5), Visit 2 (Week 10), Visit 3 (Week 15), Visit 4 (Week 20), Visit 5 (Week 30), Visit 6 (Week 40), Visit 7 (Week 55), Visit 8 (Week 75) and Study Completion Visit (Weeks 100-110).
Time Frame: Throughout Part A of the study, approximately 5 years
Population: The SAS included all participants in the enrolled population with at least one BAX 855 infusion. Number analyzed is the number of participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Main Study: On-demand: Participants age <3 years and who had not experienced two joint bleeds received on-demand treatment of 10-80IU/kg of BAX 855 IV depending on the severity of the bleeding episode.
- Part A: Main Study: Prophylaxis: Participants age <3 years or after a maximum of two joint bleeds received prophylaxis treatment with dose of 25-80 IU/kg of BAX 855 IV (based on investigator discretion) once weekly for up to 100 EDs.
Arm/Group | Part A: Main Study: On-demand | Part A: Main Study: Prophylaxis
Number analyzed (Participants) | 80 | 112
Participants
  Screening- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 75 | 40
  Screening- Binding IgG Antibodies to FVIII | 1 | 0
  Screening- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 75 | 40
  Screening- Binding IgM Antibodies to FVIII | 0 | 0
  Screening- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 75 | 40
  Screening- Binding IgG Antibodies to PEG-FVIII | 3 | 2
  Screening- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 75 | 40
  Screening- Binding IgM Antibodies to PEG-FVIII | 4 | 1
  Screening- Binding IgG Antibodies to PEG: number analyzed (Participants) | 75 | 40
  Screening- Binding IgG Antibodies to PEG | 0 | 0
  Screening- Binding IgM Antibodies to PEG: number analyzed (Participants) | 75 | 40
  Screening- Binding IgM Antibodies to PEG | 6 | 4
  Baseline- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 79 | 38
  Baseline- Binding IgG Antibodies to FVIII | 2 | 1
  Baseline- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 79 | 38
  Baseline- Binding IgM Antibodies to FVIII | 0 | 0
  Baseline- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 79 | 38
  Baseline- Binding IgG Antibodies to PEG-FVIII | 7 | 3
  Baseline- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 79 | 38
  Baseline- Binding IgM Antibodies to PEG-FVIII | 4 | 2
  Baseline- Binding IgG Antibodies to PEG: number analyzed (Participants) | 79 | 38
  Baseline- Binding IgG Antibodies to PEG | 0 | 0
  Baseline- Binding IgM Antibodies to PEG: number analyzed (Participants) | 79 | 38
  Baseline- Binding IgM Antibodies to PEG | 8 | 2
  Visit 1- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 47 | 62
  Visit 1- Binding IgG Antibodies to FVIII | 0 | 4
  Visit 1- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 47 | 62
  Visit 1- Binding IgM Antibodies to FVIII | 0 | 0
  Visit 1- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 47 | 62
  Visit 1- Binding IgG Antibodies to PEG-FVIII | 14 | 36
  Visit 1- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 47 | 62
  Visit 1- Binding IgM Antibodies to PEG-FVIII | 0 | 2
  Visit 1- Binding IgG Antibodies to PEG: number analyzed (Participants) | 47 | 62
  Visit 1- Binding IgG Antibodies to PEG | 4 | 8
  Visit 1- Binding IgM Antibodies to PEG: number analyzed (Participants) | 47 | 62
  Visit 1- Binding IgM Antibodies to PEG | 0 | 3
  Visit 2- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 20 | 76
  Visit 2- Binding IgG Antibodies to FVIII | 1 | 1
  Visit 2- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 20 | 76
  Visit 2- Binding IgM Antibodies to FVIII | 0 | 0
  Visit 2- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 20 | 76
  Visit 2- Binding IgG Antibodies to PEG-FVIII | 6 | 27
  Visit 2- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 20 | 76
  Visit 2- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Visit 2- Binding IgG Antibodies to PEG: number analyzed (Participants) | 20 | 76
  Visit 2- Binding IgG Antibodies to PEG | 2 | 3
  Visit 2- Binding IgM Antibodies to PEG: number analyzed (Participants) | 20 | 76
  Visit 2- Binding IgM Antibodies to PEG | 0 | 0
  Visit 3- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 11 | 86
  Visit 3- Binding IgG Antibodies to FVIII | 0 | 2
  Visit 3- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 11 | 86
  Visit 3- Binding IgM Antibodies to FVIII | 0 | 0
  Visit 3- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 11 | 86
  Visit 3- Binding IgG Antibodies to PEG-FVIII | 4 | 25
  Visit 3- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 11 | 86
  Visit 3- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Visit 3- Binding IgG Antibodies to PEG: number analyzed (Participants) | 11 | 86
  Visit 3- Binding IgG Antibodies to PEG | 1 | 4
  Visit 3- Binding IgM Antibodies to PEG: number analyzed (Participants) | 11 | 86
  Visit 3- Binding IgM Antibodies to PEG | 0 | 0
  Visit 4- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 5 | 87
  Visit 4- Binding IgG Antibodies to FVIII | 0 | 0
  Visit 4- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 5 | 87
  Visit 4- Binding IgM Antibodies to FVIII | 0 | 0
  Visit 4- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 5 | 87
  Visit 4- Binding IgG Antibodies to PEG-FVIII | 1 | 18
  Visit 4- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 5 | 87
  Visit 4- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Visit 4- Binding IgG Antibodies to PEG: number analyzed (Participants) | 5 | 87
  Visit 4- Binding IgG Antibodies to PEG | 0 | 1
  Visit 4- Binding IgM Antibodies to PEG: number analyzed (Participants) | 5 | 87
  Visit 4- Binding IgM Antibodies to PEG | 0 | 0
  Visit 5- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 3 | 94
  Visit 5- Binding IgG Antibodies to FVIII | 0 | 0
  Visit 5- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 3 | 94
  Visit 5- Binding IgM Antibodies to FVIII | 0 | 0
  Visit 5- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 3 | 94
  Visit 5- Binding IgG Antibodies to PEG-FVIII | 1 | 13
  Visit 5- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 3 | 94
  Visit 5- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Visit 5- Binding IgG Antibodies to PEG: number analyzed (Participants) | 3 | 94
  Visit 5- Binding IgG Antibodies to PEG | 0 | 1
  Visit 5- Binding IgM Antibodies to PEG: number analyzed (Participants) | 3 | 94
  Visit 5- Binding IgM Antibodies to PEG | 0 | 0
  Visit 6- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 1 | 94
  Visit 6- Binding IgG Antibodies to FVIII | 0 | 0
  Visit 6- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 1 | 94
  Visit 6- Binding IgM Antibodies to FVIII | 0 | 0
  Visit 6- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 94
  Visit 6- Binding IgG Antibodies to PEG-FVIII | 1 | 5
  Visit 6- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 94
  Visit 6- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Visit 6- Binding IgG Antibodies to PEG: number analyzed (Participants) | 1 | 94
  Visit 6- Binding IgG Antibodies to PEG | 0 | 0
  Visit 6- Binding IgM Antibodies to PEG: number analyzed (Participants) | 1 | 94
  Visit 6- Binding IgM Antibodies to PEG | 0 | 0
  Visit 7- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 1 | 93
  Visit 7- Binding IgG Antibodies to FVIII | 0 | 0
  Visit 7- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 1 | 93
  Visit 7- Binding IgM Antibodies to FVIII | 0 | 0
  Visit 7- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 93
  Visit 7- Binding IgG Antibodies to PEG-FVIII | 1 | 4
  Visit 7- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 93
  Visit 7- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Visit 7- Binding IgG Antibodies to PEG: number analyzed (Participants) | 1 | 93
  Visit 7- Binding IgG Antibodies to PEG | 0 | 0
  Visit 7- Binding IgM Antibodies to PEG: number analyzed (Participants) | 1 | 93
  Visit 7- Binding IgM Antibodies to PEG | 0 | 0
  Visit 8- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 1 | 90
  Visit 8- Binding IgG Antibodies to FVIII | 0 | 0
  Visit 8- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 1 | 90
  Visit 8- Binding IgM Antibodies to FVIII | 0 | 0
  Visit 8- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 90
  Visit 8- Binding IgG Antibodies to PEG-FVIII | 0 | 1
  Visit 8- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 90
  Visit 8- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Visit 8- Binding IgG Antibodies to PEG: number analyzed (Participants) | 1 | 90
  Visit 8- Binding IgG Antibodies to PEG | 0 | 0
  Visit 8- Binding IgM Antibodies to PEG: number analyzed (Participants) | 1 | 90
  Visit 8- Binding IgM Antibodies to PEG | 0 | 0
  Study Completion- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 4 | 96
  Study Completion- Binding IgG Antibodies to FVIII | 0 | 1
  Study Completion- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 4 | 96
  Study Completion- Binding IgM Antibodies to FVIII | 0 | 0
  Study Completion-Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 4 | 96
  Study Completion-Binding IgG Antibodies to PEG-FVIII | 1 | 2
  Study Completion- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 4 | 96
  Study Completion- Binding IgM Antibodies to PEG-FVIII | 1 | 0
  Study Completion- Binding IgG Antibodies to PEG: number analyzed (Participants) | 4 | 96
  Study Completion- Binding IgG Antibodies to PEG | 1 | 1
  Study Completion- Binding IgM Antibodies to PEG: number analyzed (Participants) | 4 | 96
  Study Completion- Binding IgM Antibodies to PEG | 1 | 0

4. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a participant administered an investigational product (IP) that does not necessarily have a causal relationship with the treatment. A SAE is any untoward clinical manifestation of signs, symptoms or outcomes (whether considered related to investigational product or not and at any dose) which results in death, is life-threatening, requires inpatient hospitalization, prolongation of hospitalization, is an important medical event. Number of participants with AEs and SAEs in both Part A and Part B were assessed. A participant that received on-demand treatment first and then moved to prophylaxis treatment was counted for both on-demand and prophylaxis regimens. A participant that started with prophylaxis treatment was counted only for the prophylaxis regimen even if the participant received on-demand treatment while on the prophylaxis regimen.
Time Frame: Throughout Part A and Part B of the study, approximately 9 years
Population: The SAS included all participants in the enrolled population with at least one BAX 855 infusion for Part A of the study and the IAS included all participants who received at least one FVIII inhibitor treatment with BAX 855 during the study after the date that participant moved to FVIII inhibitor treatment for Part B of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: ITI Portion (50 IU/kg Three Times Weekly Regimen): Participants received prophylaxis treatment of 50 IU/kg BAX 855 IV three times in a week.
- Part B: ITI Portion (100-200 IU/kg Daily Regimen): Participants received prophylaxis treatment of 100-200 IU/kg BAX 855 IV daily.
Arm/Group | Part A: Main Study: On-demand | Part A: Main Study: Prophylaxis | Part B: ITI Portion (50 IU/kg Three Times Weekly Regimen) | Part B: ITI Portion (100-200 IU/kg Daily Regimen)
Number analyzed (Participants) | 80 | 112 | 4 | 3
Participants
  AEs | 57 | 94 | 4 | 3
  SAEs | 18 | 35 | 1 | 3

5. Secondary Outcome: Number of Participants With At Least One Clinically Significant Changes in Vital Signs
Description: Vital signs were assessed based on body temperature, respiratory rate, blood pressure, and heart rate.
Time Frame: Throughout Part A and Part B of the study, approximately 9 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Main Study | Part B: ITI Portion
Number analyzed (Participants) | 120 | 7
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With At Least One Clinically Significant Changes in Clinical Laboratory Parameters
Description: Clinical laboratory parameters included hematology and clinical chemistry. Changes in laboratory values could be considered as AE if they were judged to be clinically significant.
Time Frame: Throughout Part A and Part B of the study, approximately 9 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Main Study | Part B: ITI Portion
Number analyzed (Participants) | 120 | 7
Participants | 53 | 1

7. Secondary Outcome: Annualized Bleeding Rate (ABR) for Prophylactic and On-demand Treatment and Immune Tolerance Induction (ITI)
Description: ABR was assessed based upon each individual bleeding episode. A bleeding episode was defined as subjective (pain consistent with a joint bleed) or objective evidence of bleeding which may or may not require treatment with FVIII. Bleeding occurring at multiple locations related to the same injury (example, knee and ankle bleed following a fall) was counted as a single bleeding episode. Mean total annualized bleed rate is reported. A participant that received on-demand treatment first and then moved to prophylaxis treatment was counted for both on-demand and prophylaxis regimens. A participant that started with prophylaxis treatment was counted only for the prophylaxis regimen even if the participant received on-demand treatment while on the prophylaxis regimen.
Time Frame: Throughout Part A and Part B of the study, approximately 9 years
Population: The SAS used for included all participants in the enrolled population with at least one BAX 855 infusion for Part A of the study and the IAS included all participants who received at least one FVIII inhibitor treatment with BAX 855 during the study after the date that participant moved to FVIII inhibitor treatment for Part B of the study.
Measure: Mean (Standard Deviation); unit: unique bleeds per year
Arm/Group | Part A: Main Study: On-demand | Part A: Main Study: Prophylaxis | Part B: ITI Portion (50 IU/kg Three Times Weekly Regimen) | Part B: ITI Portion (100-200 IU/kg Daily Regimen)
Number analyzed (Participants) | 80 | 112 | 4 | 3
unique bleeds per year | 10.004 (15.533) | 4.536 (8.657) | 7.673 (8.965) | 6.432 (14.518)

8. Secondary Outcome: Bleeding Episodes Categorized by Number of BAX 855 Infusions Required for Treatment
Description: A bleeding episode is defined as subjective (pain consistent with a joint bleed) or objective evidence of bleeding which may or may not require treatment with FVIII. The number of BAX 855 infusions needed for each bleeding episode was determined by the participant, caregiver, clinician treating the participant, and is based upon the participant's response to treatment, using the Efficacy Rating Scale for Treatment of Bleeding Episodes. Number of bleeding episodes are categorized by number of infusions required to treat the bleeding episodes. A participant that received on-demand treatment first and then moved to prophylaxis treatment was counted for both on-demand and prophylaxis regimens. A participant that started with prophylaxis treatment was counted only for the prophylaxis regimen even if the participant received on-demand treatment while on the prophylaxis regimen.
Time Frame: Throughout Part A of the study, approximately 5 years
Population: The SAS included all participants in the enrolled population with at least one BAX 855 infusion.
Measure: Number; unit: bleeding episodes
Units Other Than Participants: Number of treated bleeds
Arm/Group | Part A: Main Study: On-demand | Part A: Main Study: Prophylaxis
Number analyzed (Participants) | 80 | 112
Number analyzed (Number of treated bleeds) | 379 | 396
bleeding episodes
  Number of infusions per bleed: 0 | 7 | 14
  Number of infusions per bleed: 1 | 302 | 312
  Number of infusions per bleed: 2 | 43 | 44
  Number of infusions per bleed: 3 | 18 | 19
  Number of infusions per bleed: 4 | 4 | 1
  Number of infusions per bleed: >4 | 5 | 6

9. Secondary Outcome: Number of Bleeds by Overall Hemostatic Efficacy Rating at 24 Hours After Initiation of Treatment
Description: The participant or caregiver rated overall treatment response using a 4-point efficacy rating scale as Excellent:Full relief of pain & cessation of objective signs of bleeding after single infusion & no additional infusion is required for the control of bleeding; Good:Definite pain relief &/or improvement in signs of bleeding after single infusion & possibly requires more than 1 infusion for complete resolution; Fair:Probable &/or slight relief of pain & slight improvement in signs of bleeding after single infusion & required more than 1 infusion for complete resolution & None:No improvement or condition worsens.Number of bleeds with each efficacy rating are reported.Participant that received on-demand treatment first & then moved to prophylaxis treatment was counted for both on-demand & prophylaxis regimens.Participant that started with prophylaxis treatment was counted only for the prophylaxis regimen even if the participant received on-demand treatment while on prophylaxis regimen.
Time Frame: At 24 hours after study drug administration during Part A of the study
Population: The SAS included all participants in the enrolled population with at least one BAX 855 infusion. The number of units analyzed indicates the number of treated bleeds for which efficacy rating at 24 hours after initiation of treatment was available.
Measure: Number; unit: bleeds
Units Other Than Participants: Number of treated bleeds
Arm/Group | Part A: Main Study: On-demand | Part A: Main Study: Prophylaxis
Number analyzed (Participants) | 80 | 112
Number analyzed (Number of treated bleeds) | 158 | 184
bleeds
  Excellent | 76 | 102
  Good | 67 | 71
  Fair | 13 | 10
  None | 2 | 1

10. Secondary Outcome: Number of Bleeds by Overall Hemostatic Efficacy Rating at Bleed Resolution
Description: The participant or caregiver rated overall treatment response using a 4-point efficacy rating scale as Excellent:Full relief of pain & cessation of objective signs of bleeding after single infusion & no additional infusion is required for the control of bleeding; Good:Definite pain relief &/or improvement in signs of bleeding after a single infusion & possibly requires more than 1 infusion for complete resolution; Fair:Probable &/or slight relief of pain & slight improvement in signs of bleeding after single infusion & required more than 1 infusion for complete resolution & None:No improvement or condition worse.Number of bleeds with each efficacy rating are reported.Participant that received on-demand treatment first & then moved to prophylaxis treatment was counted for both on-demand & prophylaxis regimens.Participant that started with prophylaxis treatment was counted only for prophylaxis regimen even if the participant received on-demand treatment while on prophylaxis regimen.
Time Frame: From start of study treatment up to bleed resolution throughout Part A of the study (up to approximately 5 years)
Population: The SAS included all participants in the enrolled population with at least one BAX 855 infusion. The number of units analyzed indicates the number of treated bleeds for which overall efficacy rating was available.
Measure: Number; unit: bleeds
Units Other Than Participants: Number of treated bleeds
Arm/Group | Part A: Main Study: On-demand | Part A: Main Study: Prophylaxis
Number analyzed (Participants) | 80 | 112
Number analyzed (Number of treated bleeds) | 264 | 253
bleeds
  Excellent | 166 | 166
  Good | 83 | 77
  Fair | 12 | 9
  None | 3 | 1

11. Secondary Outcome: Weight-adjusted Consumption of BAX 855: Average Prophylactic Dose
Description: Weight-adjusted consumption of BAX 855 was determined based upon the record in participants diaries of the actual amount of BAX 855 infused as measured in the clinic. Average dose per prophylactic infusion, per month and per year are reported as categories.
Time Frame: Throughout Part A of the study, approximately 5 years
Population: The SAS included all participants in the enrolled population with at least one BAX 855 infusion. Number analyzed for each category is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Part A: Main Study: Prophylaxis
Number analyzed (Participants) | 112
IU/kg
  Average Dose [IU/kg] per Prophylactic Infusion | 45.514 (7.831)
  Average Prophylactic Dose [IU/kg] per Month: number analyzed (Participants) | 111
  Average Prophylactic Dose [IU/kg] per Month | 221.568 (85.925)
  Average Prophylactic Dose [IU/kg] per Year: number analyzed (Participants) | 83
  Average Prophylactic Dose [IU/kg] per Year | 2597.079 (783.089)

12. Secondary Outcome: Weight-adjusted Consumption of BAX 855: Average Number of Prophylactic Infusions
Description: Weight-adjusted consumption of BAX 855 was determined based upon the record in participants diaries of the actual number of BAX 855 infusions as measured in the clinic. Average number of infusions per month and year are reported as categories.
Time Frame: Throughout Part A and Part B of the study, approximately 9 years
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: infusions
Arm/Group | Part A: Main Study: Prophylaxis
Number analyzed (Participants) | 112
infusions
  Average Number of Prophylactic Infusions per Month: number analyzed (Participants) | 111
  Average Number of Prophylactic Infusions per Month | 4.900 (1.877)
  Average Number of Prophylactic Infusions per Year: number analyzed (Participants) | 83
  Average Number of Prophylactic Infusions per Year | 57.067 (16.361)

13. Secondary Outcome: Weight-adjusted Consumption of BAX 855: Average Dose
Description: Weight-adjusted consumption of BAX 855 was determined based upon the record in participants diaries of the actual amount of BAX 855 infused as measured in the clinic. Average dose to treat bleeding episode and average FVIII inhibitor treatment Dose [IU/kg] per Week, Month and per Year are reported as categories. A participant that received on-demand treatment first and then moved to prophylaxis treatment was counted for both on-demand and prophylaxis regimens. A participant that started with prophylaxis treatment was counted only for the prophylaxis regimen even if the participant received on-demand treatment while on the prophylaxis regimen.
Time Frame: Throughout Part A of the study, approximately 5 years
Population: The SAS included all participants in the enrolled population with at least one BAX 855 infusion for Part A of the study and the IAS included all participants who received at least one FVIII inhibitor treatment with BAX 855 during the study after the date that participant moved to FVIII inhibitor treatment for Part B of the study. Number analyzed for each category is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Part A: Main Study: On-demand | Part A: Main Study: Prophylaxis | Part B: ITI Portion (50 IU/kg Three Times Weekly Regimen) | Part B: ITI Portion (100-200 IU/kg Daily Regimen)
Number analyzed (Participants) | 80 | 112 | 4 | 3
IU/kg
  Average Dose [IU/kg] to Treat Bleeding Episode: number analyzed (Participants) | 80 | 112 | 0 | 0
  Average Dose [IU/kg] to Treat Bleeding Episode | 55.445 (32.826) | 63.864 (44.818) |  |
  Average FVIII Inhibitor Treatment Dose [IU/kg] per Week: number analyzed (Participants) | 0 | 0 | 2 | 3
  Average FVIII Inhibitor Treatment Dose [IU/kg] per Week |  |  | 123.510 (65.563) | 417.750 (319.694)
  Average FVIII Inhibitor Treatment Dose [IU/kg] per Month: number analyzed (Participants) | 0 | 0 | 2 | 3
  Average FVIII Inhibitor Treatment Dose [IU/kg] per Month |  |  | 537.038 (285.076) | 1816.427 (1390.068)
  Average FVIII Inhibitor Treatment Dose [IU/kg] per Year: number analyzed (Participants) | 0 | 0 | 2 | 3
  Average FVIII Inhibitor Treatment Dose [IU/kg] per Year |  |  | 6444.460 (3420.911) | 21797.128 (16680.821)

14. Secondary Outcome: Number of Participants by Hemostatic Efficacy Rating in Case of Surgery
Description: Hemostatic efficacy was assessed during & after any surgical or invasive procedures,& overall as a perioperative assessment.Operating surgeon assessed hemostatic efficacy compared to that expected for the type of procedure performed in non-hemophilic population,prior to discharge from recovery room(intraoperative),on postoperative Day 1 & at discharge or 14 days post-surgery(perioperative).Participants rated efficacy using following ratings:1.Excellent:Postoperative blood loss was ≤100% than expected;2.Good:Postoperative blood loss was up to 50% more (101-150%) than expected;3.Fair:Postoperative blood loss was more than 50% (>150%) of that expected;4.None:Significant postoperative bleeding that was result of inadequate therapeutic response despite proper dosing,necessitating rescue therapy.Perioperative ratings also considered amount of blood components required for transfusions compared to expected.Participant-provided ratings for each of the assessments are reported as categories.
Time Frame: Surgery Day 0 up to postoperative Day 14 or discharge (whichever occurs first)
Population: The Invasive Procedure Analysis Set (IPRAS) included all participants who were treated with BAX 855 for one or more surgeries or invasive procedures in the context of the study. Number of participants analyzed is the number of participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 37
Participants
  Intraoperative - Excellent: number analyzed (Participants) | 11
  Intraoperative - Excellent | 10
  Intraoperative - Good: number analyzed (Participants) | 11
  Intraoperative - Good | 0
  Intraoperative - Fair: number analyzed (Participants) | 11
  Intraoperative - Fair | 0
  Intraoperative - None: number analyzed (Participants) | 11
  Intraoperative - None | 1
  Postoperative - Excellent: number analyzed (Participants) | 11
  Postoperative - Excellent | 11
  Postoperative - Good: number analyzed (Participants) | 11
  Postoperative - Good | 0
  Postoperative - Fair: number analyzed (Participants) | 11
  Postoperative - Fair | 0
  Postoperative - None: number analyzed (Participants) | 11
  Postoperative - None | 0
  Perioperative - Excellent: number analyzed (Participants) | 11
  Perioperative - Excellent | 10
  Perioperative - Good: number analyzed (Participants) | 11
  Perioperative - Good | 0
  Perioperative - Fair: number analyzed (Participants) | 11
  Perioperative - Fair | 0
  Perioperative - None: number analyzed (Participants) | 11
  Perioperative - None | 1

15. Secondary Outcome: Blood Loss Per Participant in Case of Surgery
Description: The intraoperative blood loss was measured by determining the volume of blood and fluid removal through suction into the collection container (waste box and/or cell saver) and the estimated blood loss into swabs and towels during the procedure, per the anesthesiologist's record. Post-operatively, blood loss was determined by the drainage volume collected, which mainly consisted of drainage fluid via vacuum or gravity drain, as applicable. The assessment was done for the intra-operative time period (prior to discharge from recovery room) and for the post-operative time period (from completion of the procedure until approximately 24 hours post-surgery).
Time Frame: Surgery Day 0 up to postoperative Day 14 or discharge (whichever occurs first)
Population: The IPRAS included all participants who were treated with BAX 855 for one or more surgeries or invasive procedures in the context of the study. Number analyzed are the participants who experienced blood loss.
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | All Participants
Number analyzed (Participants) | 37
milliliters (mL)
  Observed Intra-Operative Blood Loss: number analyzed (Participants) | 17
  Observed Intra-Operative Blood Loss | 4.8 (5.43)
  Observed Post-Operative Blood Loss: number analyzed (Participants) | 0

16. Secondary Outcome: Incremental Recovery (IR) of BAX 855
Description: BAX 855 was administered in participants for the determination of FVIII IR at study site at baseline & every study visit other than study visits at 5 EDs, 15 EDs & 30 EDs. FVIII assays were done using following methods:1-stage clotting FVIII activity & FVIII chromogenic activity. Data is reported for each of these methods as categories per visit. Study Completion assessment was conducted at end of the Main Study & again at end of the ITI portion. Thus, more number of participants were analyzed at study completion visit than those who actually completed the overall study. IR is reported as a ratio of (IU/deciliter [dL])/(IU/kg), calculated as: IR = (Cmax- (C pre-infusion)) / (IU/kg), where C=concentration. Visits and their approximate time in weeks after baseline visit for individual participants: Visit 1 (Week 5), Visit 2 (Week 10), Visit 3 (Week 15), Visit 4 (Week 20), Visit 5 (Week 30), Visit 6 (Week 40), Visit 7 (Week 55), Visit 8 (Week 75) & Study Completion Visit (Weeks 100-110).
Time Frame: Baseline up to Study Completion (Up to 5 years in Part A and up to 3.5 years in Part B)
Population: The Pharmacokinetic (PK) analysis set (PKAS) included all participants in the SAS who had at least one post-dose measurement of FVIII activity without protocol deviations and/or events with potential to affect concentration (FVIII activity levels). Number analyzed is the number of participants with data available for analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | All Participants
Number analyzed (Participants) | 119
ratio
  Baseline-1-Stage Clotting: number analyzed (Participants) | 99
  Baseline-1-Stage Clotting | 1.546 (46.991)
  Baseline-Chromogenic: number analyzed (Participants) | 100
  Baseline-Chromogenic | 1.594 (55.555)
  Visit 1-1-Stage Clotting: number analyzed (Participants) | 45
  Visit 1-1-Stage Clotting | 1.452 (49.680)
  Visit 1-Chromogenic: number analyzed (Participants) | 45
  Visit 1-Chromogenic | 1.651 (43.755)
  Visit 2-1-Stage Clotting: number analyzed (Participants) | 88
  Visit 2-1-Stage Clotting | 1.345 (72.207)
  Visit 2-Chromogenic: number analyzed (Participants) | 88
  Visit 2-Chromogenic | 1.451 (57.891)
  Visit 3-1-Stage Clotting: number analyzed (Participants) | 47
  Visit 3-1-Stage Clotting | 1.439 (61.369)
  Visit 3-Chromogenic: number analyzed (Participants) | 47
  Visit 3-Chromogenic | 1.586 (54.653)
  Visit 4-1-Stage Clotting: number analyzed (Participants) | 79
  Visit 4-1-Stage Clotting | 1.558 (33.938)
  Visit 4-Chromogenic: number analyzed (Participants) | 79
  Visit 4-Chromogenic | 1.802 (31.897)
  Visit 5-1-Stage Clotting: number analyzed (Participants) | 56
  Visit 5-1-Stage Clotting | 1.588 (51.122)
  Visit 5-Chromogenic: number analyzed (Participants) | 54
  Visit 5-Chromogenic | 1.916 (28.373)
  Visit 6-1-Stage Clotting: number analyzed (Participants) | 87
  Visit 6-1-Stage Clotting | 1.714 (34.037)
  Visit 6-Chromogenic: number analyzed (Participants) | 87
  Visit 6-Chromogenic | 1.809 (46.022)
  Visit 7-1-Stage Clotting: number analyzed (Participants) | 89
  Visit 7-1-Stage Clotting | 1.742 (46.707)
  Visit 7-Chromogenic: number analyzed (Participants) | 88
  Visit 7-Chromogenic | 1.965 (20.272)
  Visit 8-1-Stage Clotting: number analyzed (Participants) | 83
  Visit 8-1-Stage Clotting | 1.634 (43.470)
  Visit 8-Chromogenic: number analyzed (Participants) | 82
  Visit 8-Chromogenic | 1.893 (36.334)
  Study Completion-1-Stage Clotting: number analyzed (Participants) | 89
  Study Completion-1-Stage Clotting | 1.819 (25.513)
  Study Completion-Chromogenic: number analyzed (Participants) | 90
  Study Completion-Chromogenic | 1.979 (23.846)
  Preoperative Assessments Surgery-1-Stage Clotting: number analyzed (Participants) | 4
  Preoperative Assessments Surgery-1-Stage Clotting | 1.481 (42.457)
  Preoperative Assessments Surgery-Chromogenic: number analyzed (Participants) | 4
  Preoperative Assessments Surgery-Chromogenic | 1.716 (45.340)

17. Secondary Outcome: Half-life (T1/2) of BAX 855
Description: The Half-life to determine FVIII half-life was an optional assessment that was planned to be performed at baseline, Visit 1, or Visit 2.
Time Frame: Pre-infusion, Post-infusion: 15-30 minutes and 24-48 hours at Baseline
Population: As pre-specified in the protocol, the determination of FVIII half-life by abbreviated PK at baseline was optional and was not performed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

18. Secondary Outcome: Immune Tolerance Induction (ITI) - Number of Participants With Partial Success and Failure of ITI
Description: Partial success defined as which meet two of following criteria, 1) inhibitor titer <0.6 BU (confirmed by a central laboratory with a second blood specimen obtained within 2 months), 2) FVIII in vivo recovery >=66% of baseline value (confirmed within a two month period), and 3) FVIII half-life >=6 hours. Failure defined as the failure to meet the criteria for partial success.
Time Frame: Up to 33 months in Part B of the study
Population: FVIII inhibitor treatment analysis set (IAS) included all participants who received at least one FVIII inhibitor treatment with BAX 855 during the study after the date that participant moved to FVIII inhibitor treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: ITI Portion
Number analyzed (Participants) | 7
Participants
  Partial Success | 1
  Failure | 1

19. Secondary Outcome: Immune Tolerance Induction (ITI) - Number of Participants With At Least One Catheter-related Complication
Description: Number of participants with catheter-related complications are reported.
Time Frame: Up to 33 months in Part B of the study
Population: IAS included all participants who received at least one FVIII inhibitor treatment with BAX 855 during the study after the date that participant moved to FVIII inhibitor treatment for Part B of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: ITI Portion (50 IU/kg Three Times Weekly Regimen) | Part B: ITI Portion (100-200 IU/kg Daily Regimen)
Number analyzed (Participants) | 4 | 3
Participants | 0 | 2

20. Secondary Outcome: Immune Tolerance Induction (ITI) - Number of Participants With Binding Immunoglobulin G (IgG) and Immunoglobulin M (IgM) Antibodies
Description: Binding IgG and IgM antibodies to Factor VIII (FVIII), Factor VIII-Polyethylene glycol (PEG-FVIII) and Polyethylene glycol (PEG) are reported as categories per visit.
Time Frame: Up to 33 months in Part B of the study
Population: The IAS included all participants who received at least one FVIII inhibitor treatment with BAX 855 during the study after the date that participant moved to FVIII inhibitor treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: ITI Portion (50 IU/kg Three Times Weekly Regimen) | Part B: ITI Portion (100-200 IU/kg Daily Regimen)
Number analyzed (Participants) | 4 | 3
Participants
  Screening- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 2 | 1
  Screening- Binding IgG Antibodies to FVIII | 0 | 1
  Screening- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 2 | 1
  Screening- Binding IgM Antibodies to FVIII | 0 | 0
  Screening- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 2 | 1
  Screening- Binding IgG Antibodies to PEG-FVIII | 0 | 1
  Screening- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 2 | 1
  Screening- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Screening- Binding IgG Antibodies to PEG: number analyzed (Participants) | 2 | 1
  Screening- Binding IgG Antibodies to PEG | 0 | 1
  Screening- Binding IgM Antibodies to PEG: number analyzed (Participants) | 2 | 1
  Screening- Binding IgM Antibodies to PEG | 0 | 0
  First Infusion- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 2 | 2
  First Infusion- Binding IgG Antibodies to FVIII | 2 | 0
  First Infusion- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 2 | 2
  First Infusion- Binding IgM Antibodies to FVIII | 0 | 0
  First Infusion- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 2 | 2
  First Infusion- Binding IgG Antibodies to PEG-FVIII | 2 | 1
  First Infusion- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 2 | 2
  First Infusion- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  First Infusion- Binding IgG Antibodies to PEG: number analyzed (Participants) | 2 | 2
  First Infusion- Binding IgG Antibodies to PEG | 0 | 0
  First Infusion- Binding IgM Antibodies to PEG: number analyzed (Participants) | 2 | 2
  First Infusion- Binding IgM Antibodies to PEG | 0 | 0
  Visit 1 (Week 2) - Binding IgG Antibodies to FVIII | 2 | 1
  Visit 1 (Week 2) - Binding IgM Antibodies to FVIII | 0 | 0
  Visit 1 (Week 2) - Binding IgG Antibodies to PEG-FVIII | 0 | 2
  Visit 1 (Week 2) - Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Visit 1 (Week 2) - Binding IgG Antibodies to PEG | 0 | 2
  Visit 1 (Week 2) - Binding IgM Antibodies to PEG | 0 | 0
  Visit 2 (Week 4) - Binding IgG Antibodies to FVIII | 1 | 1
  Visit 2 (Week 4) - Binding IgM Antibodies to FVIII | 0 | 0
  Visit 2 (Week 4) - Binding IgG Antibodies to PEG-FVIII | 1 | 1
  Visit 2 (Week 4) - Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Visit 2 (Week 4) - Binding IgG Antibodies to PEG | 0 | 0
  Visit 2 (Week 4) - Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 1- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 2 | 2
  Follow-Up Visit Month 1- Binding IgG Antibodies to FVIII | 1 | 0
  Follow-Up Visit Month 1- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 2 | 2
  Follow-Up Visit Month 1- Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 1- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 2 | 2
  Follow-Up Visit Month 1- Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 1- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 2 | 2
  Follow-Up Visit Month 1- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 1- Binding IgG Antibodies to PEG: number analyzed (Participants) | 2 | 2
  Follow-Up Visit Month 1- Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 1- Binding IgM Antibodies to PEG: number analyzed (Participants) | 2 | 2
  Follow-Up Visit Month 1- Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 2- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 2- Binding IgG Antibodies to FVIII | 1 | 0
  Follow-Up Visit Month 2- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 2- Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 2- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 2- Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 2- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 2- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 2- Binding IgG Antibodies to PEG: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 2- Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 2- Binding IgM Antibodies to PEG: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 2- Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 3- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 3- Binding IgG Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 3- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 3- Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 3- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 3- Binding IgG Antibodies to PEG-FVIII | 1 | 0
  Follow-Up Visit Month 3- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 3- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 3- Binding IgG Antibodies to PEG: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 3- Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 3- Binding IgM Antibodies to PEG: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 3- Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 4- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 3 | 2
  Follow-Up Visit Month 4- Binding IgG Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 4-Binding IgM Antibodies to FVIII: number analyzed (Participants) | 3 | 2
  Follow-Up Visit Month 4-Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 4-Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 3 | 2
  Follow-Up Visit Month 4-Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 4-Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 3 | 2
  Follow-Up Visit Month 4-Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 5- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 3 | 2
  Follow-Up Visit Month 5- Binding IgG Antibodies to FVIII | 1 | 0
  Follow-Up Visit Month 5- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 3 | 2
  Follow-Up Visit Month 5- Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 5- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 3 | 2
  Follow-Up Visit Month 5- Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 5- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 3 | 2
  Follow-Up Visit Month 5- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 5- Binding IgG Antibodies to PEG: number analyzed (Participants) | 3 | 2
  Follow-Up Visit Month 5- Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 5- Binding IgM Antibodies to PEG: number analyzed (Participants) | 3 | 2
  Follow-Up Visit Month 5- Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 6- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 6- Binding IgG Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 6- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 6- Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 6- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 6- Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 6- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 6- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 6- Binding IgG Antibodies to PEG: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 6- Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 6- Binding IgM Antibodies to PEG: number analyzed (Participants) | 4 | 2
  Follow-Up Visit Month 6- Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 7-Binding IgG Antibodies to FVIII: number analyzed (Participants) | 3 | 2
  Follow-Up Visit Month 7-Binding IgG Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 7-Binding IgM Antibodies to FVIII: number analyzed (Participants) | 3 | 2
  Follow-Up Visit Month 7-Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 7-Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 3 | 2
  Follow-Up Visit Month 7-Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 7-Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 3 | 2
  Follow-Up Visit Month 7-Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 7-Binding IgG Antibodies to PEG: number analyzed (Participants) | 3 | 2
  Follow-Up Visit Month 7-Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 7-Binding IgM Antibodies to PEG: number analyzed (Participants) | 3 | 2
  Follow-Up Visit Month 7-Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 8-Binding IgG Antibodies to FVIII: number analyzed (Participants) | 3 | 1
  Follow-Up Visit Month 8-Binding IgG Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 8-Binding IgM Antibodies to FVIII: number analyzed (Participants) | 3 | 1
  Follow-Up Visit Month 8-Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 8-Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 3 | 1
  Follow-Up Visit Month 8-Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 8-Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 3 | 1
  Follow-Up Visit Month 8-Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 8-Binding IgG Antibodies to PEG: number analyzed (Participants) | 3 | 1
  Follow-Up Visit Month 8-Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 8-Binding IgM Antibodies to PEG: number analyzed (Participants) | 3 | 1
  Follow-Up Visit Month 8-Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 9-Binding IgG Antibodies to FVIII: number analyzed (Participants) | 2 | 1
  Follow-Up Visit Month 9-Binding IgG Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 9-Binding IgM Antibodies to FVIII: number analyzed (Participants) | 2 | 1
  Follow-Up Visit Month 9-Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 9-Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 2 | 1
  Follow-Up Visit Month 9-Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 9-Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 2 | 1
  Follow-Up Visit Month 9-Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 9-Binding IgG Antibodies to PEG: number analyzed (Participants) | 2 | 1
  Follow-Up Visit Month 9-Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 9-Binding IgM Antibodies to PEG: number analyzed (Participants) | 2 | 1
  Follow-Up Visit Month 9-Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 10- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 10- Binding IgG Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 10- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 10- Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 10- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 10- Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 10- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 10- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 10- Binding IgG Antibodies to PEG: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 10- Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 10- Binding IgM Antibodies to PEG: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 10- Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 11- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 4 | 1
  Follow-Up Visit Month 11- Binding IgG Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 11- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 4 | 1
  Follow-Up Visit Month 11- Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 11- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 4 | 1
  Follow-Up Visit Month 11- Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 11- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 4 | 1
  Follow-Up Visit Month 11- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 11- Binding IgG Antibodies to PEG: number analyzed (Participants) | 4 | 1
  Follow-Up Visit Month 11- Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 11- Binding IgM Antibodies to PEG: number analyzed (Participants) | 4 | 1
  Follow-Up Visit Month 11- Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 12- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 4 | 1
  Follow-Up Visit Month 12- Binding IgG Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 12- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 4 | 1
  Follow-Up Visit Month 12- Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 12- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 4 | 1
  Follow-Up Visit Month 12- Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 12- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 4 | 1
  Follow-Up Visit Month 12- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 12- Binding IgG Antibodies to PEG: number analyzed (Participants) | 4 | 1
  Follow-Up Visit Month 12- Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 12- Binding IgM Antibodies to PEG: number analyzed (Participants) | 4 | 1
  Follow-Up Visit Month 12- Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 13- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 2 | 1
  Follow-Up Visit Month 13- Binding IgG Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 13- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 2 | 1
  Follow-Up Visit Month 13- Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 13- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 2 | 1
  Follow-Up Visit Month 13- Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 13- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 2 | 1
  Follow-Up Visit Month 13- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 13- Binding IgG Antibodies to PEG: number analyzed (Participants) | 2 | 1
  Follow-Up Visit Month 13- Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 13- Binding IgM Antibodies to PEG: number analyzed (Participants) | 2 | 1
  Follow-Up Visit Month 13- Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 14- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 14- Binding IgG Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 14- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 14- Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 14- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 14- Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 14- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 14- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 14- Binding IgG Antibodies to PEG: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 14- Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 14- Binding IgM Antibodies to PEG: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 14- Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 15- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 15- Binding IgG Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 15- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 15- Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 15- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 15- Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 15- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 15- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 15- Binding IgG Antibodies to PEG: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 15- Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 15- Binding IgM Antibodies to PEG: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 15- Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 16- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 16- Binding IgG Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 16- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 16- Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 16- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 16- Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 16- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 16- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 16- Binding IgG Antibodies to PEG: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 16- Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 16- Binding IgM Antibodies to PEG: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 16- Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 17- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 17- Binding IgG Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 17- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 17- Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 17- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 17- Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 17- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 17- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 17- Binding IgG Antibodies to PEG: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 17- Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 17- Binding IgM Antibodies to PEG: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 17- Binding IgM Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 18- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 1 | 0
  Follow-Up Visit Month 18- Binding IgG Antibodies to FVIII | 0 |
  Follow-Up Visit Month 18- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 1 | 0
  Follow-Up Visit Month 18- Binding IgM Antibodies to FVIII | 0 |
  Follow-Up Visit Month 18- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 0
  Follow-Up Visit Month 18- Binding IgG Antibodies to PEG-FVIII | 0 |
  Follow-Up Visit Month 18- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 0
  Follow-Up Visit Month 18- Binding IgM Antibodies to PEG-FVIII | 0 |
  Follow-Up Visit Month 18- Binding IgG Antibodies to PEG: number analyzed (Participants) | 1 | 0
  Follow-Up Visit Month 18- Binding IgG Antibodies to PEG | 0 |
  Follow-Up Visit Month 18- Binding IgM Antibodies to PEG: number analyzed (Participants) | 1 | 0
  Follow-Up Visit Month 18- Binding IgM Antibodies to PEG | 0 |
  Follow-Up Visit Month 19- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 19- Binding IgG Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 19- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 19- Binding IgM Antibodies to FVIII | 0 | 0
  Follow-Up Visit Month 19- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 19- Binding IgG Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 19- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 19- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  Follow-Up Visit Month 19- Binding IgG Antibodies to PEG: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 19- Binding IgG Antibodies to PEG | 0 | 0
  Follow-Up Visit Month 19- Binding IgM Antibodies to PEG: number analyzed (Participants) | 1 | 1
  Follow-Up Visit Month 19- Binding IgM Antibodies to PEG | 0 | 0
  FVIII Inhibitor Treatment Completion- Binding IgG Antibodies to FVIII: number analyzed (Participants) | 4 | 2
  FVIII Inhibitor Treatment Completion- Binding IgG Antibodies to FVIII | 0 | 0
  FVIII Inhibitor Treatment Completion- Binding IgM Antibodies to FVIII: number analyzed (Participants) | 4 | 2
  FVIII Inhibitor Treatment Completion- Binding IgM Antibodies to FVIII | 0 | 0
  FVIII Inhibitor Treatment Completion- Binding IgG Antibodies to PEG-FVIII: number analyzed (Participants) | 4 | 2
  FVIII Inhibitor Treatment Completion- Binding IgG Antibodies to PEG-FVIII | 0 | 0
  FVIII Inhibitor Treatment Completion- Binding IgM Antibodies to PEG-FVIII: number analyzed (Participants) | 4 | 2
  FVIII Inhibitor Treatment Completion- Binding IgM Antibodies to PEG-FVIII | 0 | 0
  FVIII Inhibitor Treatment Completion- Binding IgG Antibodies to PEG: number analyzed (Participants) | 4 | 2
  FVIII Inhibitor Treatment Completion- Binding IgG Antibodies to PEG | 0 | 0
  FVIII Inhibitor Treatment Completion- Binding IgM Antibodies to PEG: number analyzed (Participants) | 4 | 2
  FVIII Inhibitor Treatment Completion- Binding IgM Antibodies to PEG | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 9 years
Description: SAS:participants in enrolled population with at least 1 BAX 855 infusion.IAS:participants who received at least 1 FVIII inhibitor treatment with BAX 855 during study after participant moved to FVIII inhibitor treatment.Participant that received on-demand treatment 1st and then moved to prophylaxis treatment was counted for both on-demand & prophylaxis regimens and those who started with prophylaxis treatment was counted only for the prophylaxis regimen even if they received on-demand treatment.
Arm/Group | Part A: Main Study: On-demand | Part A: Main Study: Prophylaxis | Part B: ITI Portion (50 IU/kg Three Times Weekly Regimen) | Part B: ITI Portion (100-200 IU/kg Daily Regimen)
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/112 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 18/80 | 35/112 | 1/4 | 3/3
Other Adverse Events (participants affected / at risk) | 47/80 | 77/112 | 4/4 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Main Study: On-demand (N=80) | Part A: Main Study: Prophylaxis (N=112) | Part B: ITI Portion (50 IU/kg Three Times Weekly Regimen) (N=4) | Part B: ITI Portion (100-200 IU/kg Daily Regimen) (N=3)
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 1 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Factor VIII inhibition (Blood and lymphatic system disorders) | 5 | 6 | 0 | 1
Febrile convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 1 | 0 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 4 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 1 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Systemic viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Tongue haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 1
Vascular device occlusion (General disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Main Study: On-demand (N=80) | Part A: Main Study: Prophylaxis (N=112) | Part B: ITI Portion (50 IU/kg Three Times Weekly Regimen) (N=4) | Part B: ITI Portion (100-200 IU/kg Daily Regimen) (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bacillus test positive (Investigations) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 5 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 2 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 16 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 9 | 1 | 0
Ear infection (Infections and infestations) | 4 | 7 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 7 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 1
Influenza (Infections and infestations) | 3 | 8 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 | 6 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 18 | 2 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 5 | 7 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 6 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 17 | 31 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 1
Rhinitis (Infections and infestations) | 5 | 7 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 0 | 0
Scarlet fever (Infections and infestations) | 0 | 0 | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 12 | 27 | 2 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 1
Vessel puncture site cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 3 | 12 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 6 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT02615691/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT02615691/SAP_001.pdf